CLINICAL TRIAL: NCT04396496
Title: A Phase II Trial for the Treatment of POEMS Syndrome With Daratumumab
Brief Title: Treatment of POEMS Syndrome With Daratumumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 207442
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: POEMS Syndrome
MeSH Terms: conditions — POEMS Syndrome | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Daratumumab Injection (Experimental): Up to 12 four-week cycles of Daratumumab (DARA), in combination with the immunomodulatory drug (IMiD) lenalidomide.
  DARA is injected. Dosage calculated by weight.On Cycles 1 and 2, DARA is given on Days 1, 8,15 and 22. On Cycles 3-6,DARA is given on Days 1 and 15. On Cycles 7-12, DARA is given on Day 1.
  Lenalidomide is taken by mouth. 15 mg on Days 1-21 of each cycle.
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — DARA is a human monoclonal antibody that specifically recognizes the CD38 molecule that is expressed at a high level in a variety of hematological malignancies, including myeloma cells.
  DARA injection will be given with oral lenalidomide for up to 12 four week cycles.
  Other Names: Darzalex

SUMMARY:
This trial investigates the use of Daratumumab (DARA), an antibody directed at the human cluster of differentiation 38 (CD38) molecule, for the treatment of patients with Polyneuropathy, Organomegaly, Endocrinopathy, m Protein Component, Skin Changes (POEMS) syndrome. This trial will enroll ten subjects, who will complete 12 four-week cycles of DARA, in combination with the immunomodulatory drug (IMiD) lenalidomide. Objectives of this study include improvement in neuropathy and performance status, as well as improvement in laboratory values and survival.

DETAILED DESCRIPTION:
This trial investigates the use of DARA, an antibody directed at the human CD38 molecule, for the treatment of patients with POEMS syndrome. This trial will enroll ten subjects, who will complete 12 four-week cycles of DARA, in combination with the IMiD lenalidomide. Objectives of this study include improvement in neuropathy and performance status, as well as improvement in laboratory values and survival.

Patients will receive DARA in the outpatient setting, with infusions being administered in Infusion 4. Safety and response assessments will occur prior to Cycles 1 through 6, and at the end of DARA treatment. Once DARA is completed, response assessments are completed every 6 months for the first year, then annually until disease progression. Subjects will also be followed for overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have POEMS syndrome and meet the diagnostic criteria for POEMS syndrome as described in Appendix I.
* Both newly-diagnosed and relapsed POEMS syndrome will be eligible for inclusion.
* Patients must have a platelet count of ≥ 50,000/μL.
* Patients must be at least 18 years of age.
* Participants must have preserved renal function as defined by a serum creatinine level of < 3 mg/dL.
* Participants must have an ejection fraction by echocardiogram (ECHO) or multigated acquisition (MUGA) scan ≥ 40 percent.
* Eastern Cooperative Oncology Group ≥ 1,
* Overall Neuropathy Limitations Scale (ONLS) ≥ 1.
* Patients must have signed an institutional review board (IRB)-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the IRB.

Exclusion Criteria:

* Documented allergy to lenalidomide, DARA, mannitol, other monoclonal antibodies or human proteins and mammalian-derived products.
* Prior treatment with DARA or other CD38 monoclonal antibodies
* Patients with central nervous system (CNS) Multiple Myeloma (MM) involvement.
* Patients who have received an investigational drug or device within 4 weeks prior to enrollment or received live attenuated vaccine within 4 weeks prior to enrollment.
* Poorly controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Poor performance status will not be an exclusion criterion since POEMS patients can be expected to have significant limitations.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be accepted if the patient's life expectancy exceeds five years.
* Male and Female subjects and their partners of reproductive potential may not participate unless they have agreed to use an effective contraceptive while on study and for 3 months after cessation of DARA.
* Males who are unwilling to abstain from sperm donation while on study and for 3 months after cessation of DARA.
* Females of childbearing potential must have a negative pregnancy test documented within one week of registration.
* Females who are pregnant or nursing women may not participate.
* Patients with POEMS syndrome, who do not have disseminated bone marrow (BM) involvement and have an isolated plasmacytoma; these patients should be considered for irradiation.
* Subjects has had major surgery within 2 weeks prior to enrollment.
* Clinically significant cardiac disease, including myocardial infarction within the past 6 months or unstable or uncontrolled conditions (e.g., unstable angina or congestive heart failure) or other cardiac disease which in the opinion of the investigator would constitute a hazard for participating in the study. Some cardiac dysfunction is expected in this population.
* Participant has known chronic obstructive pulmonary disease (COPD) [defined as a forced expiratory volume in 1 second (FEV1) <50% of predicted normal, forced vital capacity (FVC), etc.] and diffusion capacity (DLCO) < 40% of predicted.), known moderate or severe persistent asthma within the last 2 years or currently has uncontrolled asthma of any classification (controlled intermittent asthma or controlled mild persistent asthma is allowed). Exception may be granted if the principal investigator documents that the patient is a candidate for therapy since alternative therapies will at least have similar or not more toxicity.
* Participant with known or suspected COPD must have an FEV1 test during screening.
* Subjects who are seropositive for human immunodeficiency virus (HIV).
* Subjects who are seropositive for hepatitis B [defined by a positive test for hepatitis B surface antigen (HBsAg)]. Subjects with resolved infection [i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen (anti-HBc)] and/or antibodies to hepatitis B surface antigen (anti-HBs) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Subjects who are seropositive for hepatitis C except in the setting of a sustained virologic response (SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab Injection: Up to 12 four-week cycles of Daratumumab (DARA), in combination with the immunomodulatory drug (IMiD) lenalidomide.
  DARA is injected. Dosage calculated by weight.On Cycles 1 and 2, DARA is given on Days 1, 8,15 and 22. On Cycles 3-6,DARA is given on Days 1 and 15. On Cycles 7-12, DARA is given on Day 1.
  Lenalidomide is taken by mouth. 15 mg on Days 1-21 of each cycle.
  Daratumumab Injection: DARA is a human monoclonal antibody that specifically recognizes the CD38 molecule that is expressed at a high level in a variety of hematological malignancies, including myeloma cells.
  DARA injection will be given with oral lenalidomide for up to 12 four week cycles.
Period: Overall Study
Arm/Group | Daratumumab Injection
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daratumumab Injection
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: There is a one-point improvement in ECOG performance score; and/or ≥ 50% reduction in ONLS score at Day 360.
Time Frame: 360 days
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab Injection
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Daratumumab Injection
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab Injection (N=2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab Injection (N=2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders, Other, specify (Skin and subcutaneous tissue disorders) | 1 (3) — hypersensitive skin, warm sensation, no flushing, no fever
Flushing (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04396496/Prot_SAP_000.pdf